CLINICAL TRIAL: NCT06297408
Title: Relma-cel for Moderate to Severe Active Systemic Lupus Erythematosus Single Arm Phase I and Phase II Randomized Controlled Open, Multicenter Study
Brief Title: Relma-cel for Moderate to Severe Active Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ming Ju Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029115
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: CD19-CART
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — relmacabtagene autoleucel; Adrenal Cortex Hormones; Immunosuppressive Agents; Biological Products

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relma-cel (Experimental): Evaluate the safety and tolerability of Relma-cel in moderate to severe active systemic lupus erythematosus (SLE) and determine the Phase II Recommended Dose (RP2D)
  Interventions: Drug: Relma-cel

INTERVENTIONS:
Drug: Relma-cel — CD19-targeted Chimeric AntigenReceptor (CAR) T Cells
  Other Names: if necessary can add other anti-SLE treatment such as corticosteroids, immunosuppressants, biologics

SUMMARY:
To assess the safety tolerability pharmacokinetics and pharmacodynamics of Relma-cel in moderate or severe active systemic lupus erythematosus (SLE) subjects in China.

DETAILED DESCRIPTION:
For phase I to evaluate the safety and tolerability of Relma-cel in moderate to severe active systemic lupus erythematosus (SLE) and determine the Phase II Recommended Dose (RP2D). For phase II to evaluation of the efficacy of Relma-cel (treatment group) in moderate to severe active SLE using the Low Disease Activity State of Lupus (LLDAS) under Phase II Recommended Dose (RP2D) compared to conventional therapy combined with or without biologics (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed an informed consent form (ICF).
2. Applicants must be between 18 and 70 years old (inclusive) at the time of signing the ICF, male or female.
3. Diagnosed with SLE according to the 2012 SLICC or 2019 EULAR/ACR version of the revised criteria.
4. Disease remaining active after receiving corticosteroids combined immunosuppressive therapy and/or biological agents, with a stable treatment plan for at least 2 months and a stable dose for at least 2 weeks before screening.

Oral corticosteroids must meet the following requirements:

1. Prednisone (or equivalent) ≥7.5 mg/day and ≤60 mg/day.
2. When used in combination with immunosuppressants, there is no minimum daily dose requirement for corticosteroids.

5. Positive antinuclear antibody, and/or anti-dsDNA antibody, and/or anti-Smith antibody at screening.

6. SELENA-2k score ≥7 points during the screening period. 7. Active organ involvement during screening period. 8. No active infection (e.g., pneumonia, tuberculosis) within 2 weeks prior to screening period.

9. Vascular access is sufficient for leukapheresis. 10. Adequate organ function:

1. Renal function: defined as creatinine clearance (Cockcroft-Gault) ≥40 mL/min calculated without hydration assistance.
2. Bone marrow function: defined as absolute neutrophil count (ANC) ≥1000 /μL, absolute lymphocyte count (ALC) ≥100 /μL, hemoglobin (Hb) ≥60 g/L, platelet count (PLT) ≥20,000 /μL. Blood transfusions and CSF must not be used to meet these requirements during the 7 days prior to eligibility screening.
3. Liver function: defined as alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN, total bilirubin < 2.0 mg/dL (total bilirubin < 3.0 mg/dL in subjects with Gilbert syndrome, except for caused by SLE).
4. Coagulation function: defined as international ratio (INR) or activated partial thromboplastin time (APTT) ≤1.5×ULN.
5. Lung function: defined as ≤CTCAE grade 1 dyspnea and blood oxygen saturation (SpO2) ≥92% in indoor air (measured by pulse oximeter).
6. Cardiac function: defined as left ventricular ejection fraction (LVEF) ≥40% as assessed by echocardiography (ECHO) or cardiac radionuclide angiography (MUGA) within 8 weeks prior to screening.

11. Fertile women (defined as all women biologically capable of becoming pregnant) must consent to the use of a highly effective contraceptive method for contraception from at least 28 days before the start of lymphodepleting and 2 years after infusion of Relma-cel (including the duration of the dose-interrupted study treatment). Men whose partners are fertile must agree to use an effective barrier method of contraception from the start of lymphodepleting until 2 year after Relma-cel infusion and should not donate semen or sperm throughout the study period.

12. Fertile women must test negative for serum beta human chorionic gonadotropin (β-hCG) at the time of screening and within 48 hours before the first day of lymphodepleting treatment.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria should not be included in this study

1. Severe lupus nephritis within 2 months before screening requires hemodialysis, or treatment with prednisone(or equivalent hormone) ≥100 mg/d for more than 14 days.
2. Suffering from lupus crisis within 1 months before screening, assessed by the researcher as unsuitable for participation in this study.
3. Clinically significant central nervous system diseases or pathological changes not caused by lupus prior to screening, including but not limited to: cerebrovascular accident, aneurysm, epilepsy, convulsions/convulsions, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis. Central nervous system manifestations caused by lupus before screening, including but not limited to lupus headache, epileptic seizures, cognitive impairment, impaired intellectual function, visual impairment, etc.
4. Combined with other autoimmune diseases, systemic treatment is required.
5. History of major organ transplantation (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
6. When screening:

1) Active hepatitis B. However, hepatitis B surface antigen (HBsAg) positive and/or anti-hepatitis B core antibody (HBcAb) positive, and HBV DNA below the lower limit of the central reference value are eligible for inclusion in this study, and investigators need to provide preventive antiviral therapy to participants as appropriate.

2) Hepatitis C or human immunodeficiency virus (HIV) or syphilis infection. 7. A history of any of the following cardiovascular diseases in the 6 months prior to screening: Class III or IV heart failure as defined by the New York Heart Association (NYHA), myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmia, any ventricular arrhythmia, or other clinically significant heart disease.

8. Use any other clinical study drugs within 1 month before screening. However, if the research treatment is ineffective or the disease relapses, and at least 3 half-life period have been passed before screening, enrollment is allowed.

9. Previously received CAR-T cell or other genetically modified T cell therapies.

10. There was a history of ≥grade 2 bleeding within 30 days prior to screening, or long-term treatment with anticoagulants (such as warfarin, low molecular weight heparin, or factor Xa inhibitors).

11. Plasma exchange, plasma separation or hemodialysis were performed within 14 days before leukapheresis.

12. Use any live vaccine against infectious diseases within 1 month prior to screening.

13. Known life-threatening allergic reactions, hypersensitivities, or intolerances to Relma-cel or their excipients, including DMSO.

14. A history or evidence of suicidal thoughts in the 6 months before signing the ICF, or any suicidal behavior in the 12 months prior, or is considered by the investigator there is a significant risk of suicide.

15. Malignant tumor within 2 years before signing the ICF. Exceptions include non-melanoma skin cancer after radical treatment, localized prostate cancer, biopsy-confirmed cervical carcinoma in situ or squamous intraepithelial lesions detected by cervical smear, and completely resected breast carcinoma in situ.

16. Pregnant or lactating women. 17. Other situations in which the investigator determines that the subject has poor compliance or is unwilling or unable to comply with the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
DLT rate | 6months
  The incidence of dose-limiting toxicity
determine RP2D | 6months
  To determine RP2D(Phase 2 recommended dose)

SECONDARY OUTCOMES:
SELENA-SLEDAI | 3 months after CD19 cCAR T cells infusion
  0 to 4 is basically no disease activity;5 to 9 is light activity;10 to 14 is moderate activity;≥15 is considered heavy activity.
BILAG -2004 | 3 months after CD19 cCAR T cells infusion
  The BILAG 2004 index categorizes disease activity into 5 different levels from A-E.Grade A represents very active disease.
PGA (physician global assessment) score | 3 months after CD19 cCAR T cells infusion
  The PGA scale ranges from "no disease activity" (0) to the "most severe disease activity" (3).the score is between 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: xiaofeng zeng, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mackensen A, Muller F, Mougiakakos D, Boltz S, Wilhelm A, Aigner M, Volkl S, Simon D, Kleyer A, Munoz L, Kretschmann S, Kharboutli S, Gary R, Reimann H, Rosler W, Uderhardt S, Bang H, Herrmann M, Ekici AB, Buettner C, Habenicht KM, Winkler TH, Kronke G, Schett G. Anti-CD19 CAR T cell therapy for refractory systemic lupus erythematosus. Nat Med. 2022 Oct;28(10):2124-2132. doi: 10.1038/s41591-022-02017-5. Epub 2022 Sep 15. PMID 36109639